CLINICAL TRIAL: NCT04504019
Title: Clinical Outcomes of Carpal Tunnel Release With and Without Ultrasound Guidance
Brief Title: Clinical Outcomes of USCTR vs. mOCTR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WRNMMC-2020-0278
Record Dates: First submitted 2020-06-22; First posted 2020-08-07 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Carpal Tunnel
Keywords: Median Nerve Neuropathy Treatments; Ultrasound Guided Carpal Tunnel Release (USCTR); Military; Minimally Invasive Carpal Tunnel Release
MeSH Terms: conditions — Median Neuropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- USCTR Procedure (Experimental): Participants will undergo the USCTR procedure with SX-One MicroKnife®, also known as UltraGuideCTR
  Interventions: Device: USCTR
- mOCTR Procedure (Active Comparator): Participants will undergo the traditional mOCTR procedure.
  Interventions: Procedure: mOCTR

INTERVENTIONS:
Device: USCTR — Ultrasound guided CTR via a single < 1 cm wrist or palmar incision. The procedure will be performed using the SX-One MicroKnife®, also known as UltraGuideCTR
  Arms: USCTR Procedure
Procedure: mOCTR — Mini-open CTR via a single 1-3cm palmar incision
  Arms: mOCTR Procedure

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common peripheral entrapment neuropathy and affects 3-6% of adults in the United States. In patients with severe or refractory symptoms, carpal tunnel release (CTR) represents the definitive management option, and over 550,000 CTRs are performed annually in the United States with over 90% of patients reporting clinical improvement. Currently available CTR techniques include mini-open CTR via a single, 1-3 cm palmar incision (mOCTR), endoscopic CTR via one (wrist) or two (wrist and palm) 1-2 cm incisions (ECTR), and ultrasound guided CTR via a single < 1 cm wrist or palmar incision (USCTR or CTR-US). The primary objective is to assess the impact of USCTR vs mOCTR in a military population. Investigators hypothesize that USCTR using the SX-One MicroKnife, also known as UltraGuideCTR, will safely and non-inferiorly improve symptoms of carpal tunnel syndrome compared to traditional mOCTR, without greater less loss of military duty days. This study is a single-site randomized controlled trial.

Participants with CTS will be randomized to a study arm and receive treatment with USCTR vs. traditional mOCTR. All patients will be followed for a period of 24 months with respect to standard clinical data, military relevant data, and validated patient related outcome measures (PROMs). Data will be collected at 1 week, 2 weeks, 3 weeks, 1 month, 6 weeks, 3 months, 6 months, and 12 months, and 24 months post-CTR procedure, with the primary focus being on outcomes up to 1 year.

DETAILED DESCRIPTION:
Clinical outcomes of up to 83 participants (updated target sample size) treated with USCTR vs. traditional mOCTR will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Adults age ≥18 years
* DEERS Eligible
* Fluent in speaking, reading, and understanding English
* Clinical diagnosis of Carpal Tunnel Syndrome (CTS)
* Candidate for surgical CTR based on severe and/or refractory symptoms
* Confirmatory electrodiagnostic test indicating median neuropathy at the wrist (abnormal findings)
* Ultrasound findings consistent with median nerve enlargement in the carpal tunnel

Exclusion Criteria:

* Previous carpal tunnel release or previous wrist surgery on the ipsilateral side
* Carpal tunnel injection with corticosteroid within 6 weeks prior to anticipated study procedure
* Previous traumatic injury to the median nerve or any of its branches on the ipsilateral side
* History of medical condition that would preclude safe participation in study procedures (e. g. complex regional pain syndrome (CRPS), upper limb vascular disease (including thoracic outlet syndrome), Raynaud's phenomenon, etc.)
* Inability to stop anticoagulation medications (Plavix, Coumadin/Warfarin, Xarelto), or unable to be bridged with Lovenox
* Unable to understand and provide written informed consent
* Contraindication to proceeding with USCTR based on diagnostic ultrasound (i.e. identification of anomalous anatomic structures such as transligamentous thenar motor branch or space occupying lesions within the carpal tunnel)
* Electrodiagnostic evaluation of the carpal tunnel which indicates normal findings

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2025-08-06 (Actual)

PRIMARY OUTCOMES:
Measure the effect of USCTR vs mOCTR on the longitudinal change in QuickDASH. | Change from baseline to 1 week, 2 weeks, 3 weeks, 1 month, 6 weeks, 3 months, 6 months, 12 months, and 24 months post CTR procedure
  QuickDash is a region-specific PROM consisting of 11 items measuring the difficulty in performing physical activities relevant to shoulder, arm or hand function. Each item is scored on a scale of 1-5 and a final score of 0 to 100 is calculated, with higher scores representing greater degrees of upper extremity disability (0 points indicate no disability and 100 points indicates maximum disability).
  For the primary analysis, change in QuickDASH score will be tracked across the first five occasions of assessment (i.e. baseline - 1 month) and the patient-level average trend will be compared between randomized groups. As a secondary analysis, change in QuickDASH will be tracked over the full duration of follow-up, with the primary focus being on outcomes up to 1 year.
Measure the effect of USCTR vs mOCTR on the longitudinal change in BCTQ-SSS. | Change from baseline to 1 week, 2 weeks, 3 weeks, 1 month, 6 weeks, 3 months, 6 months, 12 months, and 24 months post CTR procedure
  The BCTQ is a PROM for CTS and is the most commonly used outcome measure for CTS. Each item on the 11-item symptom severity scale (BCTQ-SSS) is graded from 1 (mildest) to 5 (most severe). Outcomes are typically recorded as a mean score.
  For the primary analysis, change in BCTQ-SSS score will be tracked across the first five occasions of assessment (i.e. baseline - 1 month) and the patient-level average trend will be compared between randomized groups. As a secondary analysis, change in BCTQ-SSS will be tracked over the full duration of follow-up, with the primary focus being on outcomes up to 1 year.
Measure the effect of USCTR vs mOCTR on the longitudinal change in hand grip strength. | Change from baseline to 3 months, and 12 months post CTR procedure
  Manually tested using a handheld dynamometer.
  Between the mOCTR and USCTR groups, will compare hand grip strength across each time point (i.e. baseline - 3 months; baseline - 12 months).
Measure the effect of USCTR vs mOCTR on the longitudinal change in pinch (tip, palmar, and key) strength. | Change from baseline to 3 months, and 12 months post CTR procedure
  Manually tested using a pinch gauge.
  Between the mOCTR and USCTR groups, will compare pinch (tip, palmar, and key) strength across each time point (i.e. baseline - 3 months; baseline - 12 months).
Measure the impact of USCTR vs mOCTR on participant perception of change in overall physical condition | Change from 1 week to 2 weeks, 3 weeks, 1 month, 6 weeks, 3 months, 6 months, 12 months, and 24 months post CTR procedure
  Participant self reported change in physical condition. Participant will select one response from the following descriptions to rate overall condition from the time they began treatment to the designated time-point: A very great deal worse; About the same; A very great deal better; A great deal worse; A great deal better; Quite a bit worse; Quite a bit better; Moderately worse; Moderately better; Somewhat worse; Somewhat better; A little bit worse; A little bit better; A tiny bit worse(almost the same); A tiny bit better (almost the same)
  The Global Rate of Change Scale (GROC) will be captured at nine occasions of assessment: baseline and 1 week, 2 weeks, 3 weeks, 1 month, 6 weeks, 3 months, 6 months, 12 months, and 24 months post-CTR. The primary focus will be on outcomes up to 1 year.
Change in military work status as assessed using single-item self-report assessment | Captured at 1 week, 2 weeks, 3 weeks, 1 month, 6 weeks, 3 months, 6 months, 12 months, and 24 months post CTR procedure
  Participants will complete a questionnaire to depict when normal work or daily activities commenced.
  The primary focus will be on outcomes up to 1 year.
Surgical time during procedure (minutes) | At time of procedure, measured as day 0
  On the day the participant receives their study assigned procedure (USCTR vs. mOCTR), clinical team will record surgical time to perform the procedure in minutes
Change in self-reported satisfaction as assessed using a satisfaction rating scale | Captured at 1 week, 2 weeks, 3 weeks, 1 month, 6 weeks, 3 months, 6 months, 12 months, and 24 months post CTR procedure
  Participants will rate satisfaction with the following: completely dissatisfied, mostly dissatisfied, somewhat satisfied, neither satisfied or dissatisfied, somewhat satisfied, mostly satisfied, or completely satisfied.
  Completely dissatisfied with represent the lowest score, and completely satisfied will represent the highest score.
  Will compare participant satisfaction across arms in terms of symptom improvement, incision appearance, and recovery, with the primary focus being on outcomes up to 1 year.
Change in self-reported pain as assessed using the 11-item Numeric Pain Rating Scale (NPRS) participant pain levels over 1 month following the CTR procedure. | Captured at 1 week, 2 weeks, 3 weeks, and 1 month post CTR procedure
  The 11-item NPRS scale is a unidimensional measure of pain intensity. It is a segmented numeric version of the visual analog scale in which participants will select a whole number (0-10 integers) that best reflects the intensity of their pain. The scale ranges from '0' representing one pain extreme (e.g. no pain) to '10' representing the other pain extreme (e.g. worst possible pain).
Change in pain medication usage as assessed using single-item self-report assessment | Captured at 1 week, 2 weeks, 3 weeks, 1 month, 6 weeks, 3 months, 6 months, 12 months, and 24 months post CTR procedure
  Participant self-reported pain medication usage. Participant will respond with responses ranging from "less than once a week', "once a week", "several times a week", "daily", "multiple times per day", "or did not use". "Did not use" will represent the minimum value, and "multiple times per day" will represent the maximum value.
  Participant self-reported pain medication usage (e.g., cumulative dosage, drug category, duration of use, etc.) will be captured at nine occasions of assessment: 1 week, 2 weeks, 3 weeks, 1 month, 6 weeks, 3 months, 6 months, 12 months, and 24 months post-CTR. The primary focus will be on outcomes up to 1 year.
Incision length in cm | At time of procedure, measured as day 0
  On the day the participant receives their study assigned procedure (USCTR vs. mOCTR), clinical team will record incision length in cm
Change in self-reported pain as assessed using the 11-item Numeric Pain Rating Scale (NPRS) | At time of procedure, measured as day 0
  Using the 11-item Numeric Pain Rating Scale (NPRS), compare the distributions of participant self-reported pain at both pre- and immediately -post CTR procedure between the USCTR and mOCTR groups.
  The 11-item NPRS scale is a unidimensional measure of pain intensity. It is a segmented numeric version of the visual analog scale in which participants will select a whole number (0-10 integers) that best reflects the intensity of their pain. The scale ranges from '0' representing one pain extreme (e.g. no pain) to '10' representing the other pain extreme (e.g. worst possible pain).
Change in self-reported pain as assessed using the modified 2-item CTS Palmar Pain Scale (4 items) over 1 month following CTR procedure | Captured at 1 week, 2 weeks, 3 weeks, and 1 month post CTR procedure
  The modified 2-item CTS Palmar Pain Scale (4 items on palmar and incision pain) inquires about severity of pain. Each item has five-six possible response options which range from 1 (no pain) to 5/6 (very severe). The symptom score is the mean of all answered items; higher scores indicate worse symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Miller, MD, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-12-19): https://cdn.clinicaltrials.gov/large-docs/19/NCT04504019/ICF_000.pdf